CLINICAL TRIAL: NCT06071741
Title: The Percutaneous Coronary Intervention Registry in University Medical Center of Ho Chi Minh City
Acronym: UMC-PCI
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 257/2023/HD-DHYD
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Registry; Vietnam; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCI group: Patients undergoing Percutaneous Coronary Intervention
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — balloon angioplasty, stent implantation, atherectomy, intravascular ultrasound.

SUMMARY:
* This is a hospital-based registry study that will be to describe clinical and paraclinical features, procedural-related characteristics, short and long-term outcomes, hospital costs of patients undergoing percutaneous coronary intervention (PCI) at University Medical Center of Ho Chi Minh City (UMC), together with investigating predictors for patients' adverse clinical outcomes.
* The specific objectives of this study are:

  * To validate a framework/model of PCI registry in UMC
  * To investigate the demographic, clinical of cardiovascular diseases and procedural characteristics of patient undergoing PCI in UMC
  * To investigate the procedural success, in-hospital adverse events and patient outcomes at one-month, three-month, twelve-month, three-year and five-year follow-up after PCI in UMC
  * To estimate in-hospital and procedural costs associated with PCI in UMC
  * To develop a prognostic prediction model for patients after PCI in UMC

DETAILED DESCRIPTION:
* The central single-center registry study will be conducted and monitored over a period of 5 years on patients who have undergone percutaneous coronary intervention (PCI) at UMC. The UMC-PCI registry study will utilize the ACS-PCI variables that have been standardized by EUROHEART.
* This study will help to understand the practice of PCI in one of the biggest PCI centers in Southern Vietnam, as it assesses the characteristics, treatments and outcomes of CVD patients who receive PCI procedures, as well as information regarding PCI cost. The collection tools capture the data that measures adherence to validated EUROHEART's data set about ACS-PCI.
* Through the capture and reporting of trusted and reliable data, UMC-PCI Registry helps participants measure and benchmark in specific aims:
* To examine patient baseline characteristics by demographics, medical history, clinical manifestations before PCI
* To obtain information of revascularization procedure with: coronary balloon, drug-eluting balloon, bare-metal stent, drug-eluting stent, bioresorbable vascular scaffold, rotational atherectomy device, directional coronary atherectomy device, thrombus aspiration, distal protection, the use of mechanical circulatory support devices, procedural success/failure and access site
* To estimate successful rate in procedure performance and clinical appearance
* To investigate peri-procedure and in-hospital complications
* To obtain results of cardiac enzymes and other biomarkers after procedure
* To examine discharge medication and follow-up plan
* To obtain: MACE (Major Adverse Cardiac Event), patient symptoms, wellbeing, medications and laboratory results at the one-month, three-month, twelve-month, three-year and five-year follow-up. The trial will be conducted in the University Medical Center at Ho Chi Minh City. The Interventional Cardiology department at Ho Chi Minh City is the setting to recruit patients requiring PCI in Ho Chi Minh City as well as neighboring provinces. Approximately 1200 cases are performed annually in this department. This is a relatively large number and has the potential to conduct meaningful studies regarding this field.
* All patients with coronary artery diseases with PCI agreeing to participate will be included. Patients' data will be collected and managed through REDCap. These data include information of patients' demographics, clinical history and presentations, treatments, and blood test results. The data collection forms are based on EUROHEART's data set.
* After PCI, data related to the procedure are collected including indications for performing the procedure, coronary angiogram result, degree of stenosis, coronary blood flow grade, thrombus burden, type, number and total length of stent(s) used, the usage of advance techniques during the procedure (e.g., use of intravascular ultrasound, measures of fractional flow reserve, and use of rotational atherectomy). These data will detail how PCI is performed, both in terms of technical aspects and patient outcomes.
* In-hospital complications, discharge medications, intervention costs, such as angiography procedure costs, balloon and stent expense, and additional supporting devices charges..., as well as overall in-hospital costs will be gathered. These will help monitoring procedure's complications, identifying factors influencing the occurrence of these events, optimization of post-procedural medications and giving an overall view of the economic burden faced by the patient and the healthcare system.
* All patients will be contacted by phone after one-month, three-month, twelve-month, three-year and five-year following the PCI procedure. The investigators will collect information on patients' status and incident data on MACE, bleeding complication, medications and impact of angina on quality of life using SAQ-7.
* The data will be entered into the REDCap program, which will subsequently be processed with the R 4.1.0 program. With a p value < 0.05 and a 95 percent confidence interval, all of the analyses are statistically significant. The investigators employ descriptive statistics, one-variable statistics, and statistics with multiple variables. Qualitative data will be presented as rates and percentages using descriptive statistics, the data will then be processed using the Chi-square test. The investigators report quantitative data as mean (standard deviation) for normal distributions and median (interquartile range) for other distributions. The investigators will use an unpaired t-test to compare means.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing any PCI procedure(s) in given timeframe will be included in this registry

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients performing any PCI procedure(s) in given timeframe will be included in this registry
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
MACE endpoint (Major adverse cardiovascular event) | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Composite endpoint (MACE: major adverse cardiovascular event): occurence of cardiovascular death, non-fatal or fatal myocardial infraction, non-fatal or fatal stroke, Target Lesion revascularisation or Target Vessel Revascularisation

SECONDARY OUTCOMES:
Rate of Ischemia driven target lesion revascularization (ID-TLR) | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Ischemia driven target lesion revascularization (ID-TLR)
Rate of Target Lesion Revascularization (TLR) | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  All Target Lesion Revascularization
Rate of Target Vessel Revascularization (TVR) | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  All Target Vessel Revascularization
Rate of Ischemia driven target vessel revascularization (ID-TVR) | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Ischemia driven target vessel revascularization (ID-TVR)
Rate of Ischemia driven non target vessel revascularization (ID-NTVR) | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Ischemia driven non target vessel revascularization (ID-NTVR)
Rate of All revascularization | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  All revascularization
Rate of Death | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Cardiovascular Death, All-Cause Death
Composite: Cardiovascular death or myocardial infarction | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Composite: Cardiovascular death or myocardial infarction
Composite: All-cause death or myocardial infarction | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Composite: All-cause death or myocardial infarction
Composite: All-cause death, myocardial infarction or target vessel revascularization | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Composite: All-cause death, myocardial infarction or target vessel revascularization
Anginal Status | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Anginal Status by Seattle Angina Questionnaire-7 (SAQ-7)
Rate of Stent Thrombosis | Time-To-Event measure up to 5-year from baseline: 1-month, 3-month, 12-month, 3-year, 5-year follow-up
  Composite: Probable or definite stent thrombosis Probable Stent Thrombosis Definite Stent Thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided